CLINICAL TRIAL: NCT03168867
Title: Effectiveness Trial of an E-Health Intervention To Support Diabetes Care in Minority Youth (3Ms)
Acronym: 3Ms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Deborah Ellis, Ph.D., Professor of Family Medicine and Public Health Sciences Wayne State University School of Medicine, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 015117B3E; R01DK110075 (NIH); 1R01DK110075-01A1 (NIH)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: insulin dependent diabetes mellitus; adolescents/young adults; e-health intervention; parental monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Educational Control (No Intervention): Participants in the standard educational control group will be provided with standard care regarding type 1 diabetes management during their routine clinic visits as usual. The standard care will be consistent with diabetes education provided by each of the study sites.
- The 3Ms Intervention + Standard Care (Experimental): Parents will complete the first intervention session in the diabetes clinic immediately after baseline data collection and randomization. The subsequent two intervention sessions will also be conducted during regularly scheduled diabetes clinic visits.
  Interventions: Behavioral: The 3Ms Intervention

INTERVENTIONS:
Behavioral: The 3Ms Intervention — The 3 Ms is a brief e-health intervention delivered via an internet-based software application (CIAS) that incorporates principles of Motivational Interviewing. The goal of the 3 Ms intervention is to increase caregiver motivation to supervise children's daily diabetes care. The intervention consists of 3 brief sessions that are delivered at routine diabetes clinic appointments.
  Arms: The 3Ms Intervention + Standard Care

SUMMARY:
The purpose of the study is to conduct a multicenter, randomized effectiveness trial of The 3Ms. The proposed study will use an effectiveness-implementation "Hybrid 1" design. In this design, the primary goal is to determine whether an intervention works in a real-world setting, but the design also answers secondary questions such as the relationship between treatment dose and treatment outcome and what factors affect the actual delivery of the intervention in the clinics (staff burden, workflow interference etc).

DETAILED DESCRIPTION:
The study will be conducted at 3 clinics in the Detroit area (Children's Hospital of Michigan (CHM); Ascension St. John Children's Hospital; William Beaumont Children's Hospital) and 4 clinics in the Chicago area. Wayne State University (WSU) will function as the coordinating center for the trial and will be responsible for overseeing the adequacy all aspects of trial management, including recruitment, retention, data collection, data management and statistical analyses. 212 African American (AA) adolescents with type 1 diabetes and their primary caregivers will be enrolled across all sites (half will be enrolled at WSU and half at the 4 Chicago sites). Families will be randomized to one of two arms: The 3Ms intervention (parental motivation for supervision of adolescent DSM) or standard educational control. In the 3Ms condition, parents will receive a brief (10-20 minute) computer delivered intervention at three consecutive routine diabetes clinic visits that is designed to increase parental motivation to supervise adolescent diabetes management. In the control condition, parents will receive computer-delivered education materials regarding type 1 diabetes. Data collection will be completed in the diabetes clinic at baseline and then at 6, 12 and 18 months after baseline in the families' home. Data collection is completed by the adolescent and caregiver on a tablet computer and includes questionnaires to assess adolescent diabetes management, parental supervision of diabetes management, family relationships and youth quality of life. Blood will also be collected to measure HbA1c (mean blood glucose level). Medical record data will also be collected. The data analyses will be intent-to-treat, meaning that all randomized participants are included regardless of the intervention dose received. Trial data will analyzed using the linear mixed effect model (LME) for repeated measures.

In addition to the clinical trial, 20 diabetes clinic staff members (5 at WSU from the CHM clinic; 15 from the Chicago clinics) will also be recruited to participate in qualitative interviews upon completion of the trial. The purpose of the interview is to identify barriers and facilitators of use of the 3Ms intervention at the level of the individual clinician, the diabetes clinic and the organization (hospital). Interviews will be audiotaped and subsequently transcribed for coding.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10 years 0 months - 15 years, 11 months
* Diagnosed with Type 1 diabetes
* Diagnosed for at least 6 months
* African American
* Residence within 30 miles of a recruitment site (Children's Hospital of Michigan, Ann and Robert H. Lurie Children's Hospital of Chicago, Children's Hospital University of Illinois, or La Rabida Children's Hospital of Chicago)
* Primary caregiver willing to participate

Exclusion Criteria:

* Mental health conditions that might compromise data integrity (e.g., developmental delay, schizophrenia, psychosis, current suicidality, homicidality)
* Co-morbid medical condition resulting in atypical diabetes management (e.g., cystic fibrosis)
* Inability to speak or read English
* Child is in out-of-home placement

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Ellis, Ph.D., Principal Investigator — Wayne State University
Locations (7):
- United States (7):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital University of Illinois, Chicago, Illinois
  - UChicago Medicine Comer Children's Hospital, Chicago, Illinois
  - La Rabida Children's Hospital, Chicago, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - Ascension St. John Children's Hospital, Detroit, Michigan
  - William Beaumont Children's Hospital, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knauft KM, Jacques-Tiura AJ, Carcone AI, Evans MA, Weissberg-Benchell J, Buggs-Saxton C, Boucher-Berry C, Miller JL, Drossos T, Dekelbab MB, Ellis D. Blood Glucose Levels and Diabetes Family Conflict in Black Adolescents with Type 1 Diabetes During the COVID-19 Pandemic. Behav Med. 2025 Aug 27:1-15. doi: 10.1080/08964289.2025.2543265. Online ahead of print. PMID 40859913
- [Derived] Knauft KM, Jacques-Tiura AJ, Idalski Carcone A, Evans M, Weissberg-Benchell J, Buggs-Saxton C, Boucher-Berry C, Miller JL, Drossos T, Dekelbab B, Ellis DA. The moderating role of diabetes distress on the effect of a randomized eHealth intervention on glycemic control in Black adolescents with type 1 diabetes. J Pediatr Psychol. 2024 Aug 1;49(8):538-546. doi: 10.1093/jpepsy/jsae033. PMID 38775162
- [Derived] Ellis D, Carcone AI, Templin T, Evans M, Weissberg-Benchell J, Buggs-Saxton C, Boucher-Berry C, Miller JL, Drossos T, Dekelbab MB. Moderating Effect of Depression on Glycemic Control in an eHealth Intervention Among Black Youth With Type 1 Diabetes: Findings From a Multicenter Randomized Controlled Trial. JMIR Diabetes. 2024 Apr 9;9:e55165. doi: 10.2196/55165. PMID 38593428

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Educational Care Control: Participants in the standard educational control group received education regarding type 1 diabetes management during their routine clinic visits. Education was consistent with the standard care provided by each of the study sites.
- The 3Ms Intervention + Standard Educational Care: The 3Ms was a brief e-health intervention delivered via an internet-based software application (CIAS) that incorporated principles of Motivational Interviewing. The goal of The 3Ms was to provide psychoeducation regarding the value of daily parental supervision of adolescent diabetes management and increase the primary caregiver's motivation to supervise adolescents' daily diabetes management. The intervention consisted of three brief 10-15 minute sessions delivered on a tablet computer during routine diabetes clinic appointments.
Period: Overall Study
Arm/Group | Standard Educational Care Control | The 3Ms Intervention + Standard Educational Care
Started | 74 | 75
Completed | 73 | 70
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Educational Care Control | The 3Ms Intervention + Standard Educational Care | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (1.5) | 13.1 (1.8) | 13.4 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 46 | 86
  Male | 34 | 29 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 74 | 75 | 149
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 11.5 (2.8) | 11.5 (2.7) | 11.5 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control
Description: Hemoglobin A1c (HbA1c)
Time Frame: Baseline, 6, 13 and 18 month follow-up
Population: The analyses were intent-to-treat. All randomized participants were included in the analyses
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Standard Educational Care Control | The 3Ms Intervention + Standard Educational Care
Number analyzed (Participants) | 74 | 75
percentage of glycosylated hemoglobin
  Baseline | 11.51 (2.8) | 11.48 (2.7)
  6 month follow-up: number analyzed (Participants) | 70 | 72
  6 month follow-up | 11.55 (2.7) | 11.14 (2.6)
  13 month follow-up: number analyzed (Participants) | 67 | 68
  13 month follow-up | 11.47 (2.9) | 11.09 (2.7)
  18 month follow-up: number analyzed (Participants) | 62 | 59
  18 month follow-up | 11.47 (2.9) | 10.76 (2.5)
Statistical Analysis 1: Comparison: Standard Educational Care Control vs The 3Ms Intervention + Standard Educational Care; Test type: Superiority; p < .05, Mixed Models Analysis

2. Secondary Outcome: Regimen Adherence (Objective)
Description: Glucose Meter (frequency of testing)
Time Frame: Baseline, 6 months, 13 months, and 18 months
Reporting Status: Not Posted

3. Secondary Outcome: Diabetes Management (Self-reported)
Description: Diabetes Management Scale (DMS)
Time Frame: Baseline, 6 months, 13 months, and 18 months
Reporting Status: Not Posted

4. Secondary Outcome: Parental Monitoring of Diabetes Care (Self-reported)
Description: The Parental Monitoring of Diabetes Care-Revised (PMDC-R)
Time Frame: Baseline, 6 months, 13 months, and 18 months
Reporting Status: Not Posted

5. Secondary Outcome: Diabetes- Specific Family Functioning (Self-reported)
Description: Diabetes Family Conflict Scale (DFCS-R)
Time Frame: Baseline, 6 months, 13 months, and 18 months
Reporting Status: Not Posted

6. Secondary Outcome: Adolescent Depression (Self-reported)
Description: Patient Reported Outcomes Measurement Information System (PROMIS)
Time Frame: Baseline, 6 months, 13 months, and 18 months
Reporting Status: Not Posted

7. Secondary Outcome: Executive Functioning (Self-reported)
Description: Behavior Rating Inventory of Executive Function (BRIEF)
Time Frame: Baseline, 6 months, 13 months, and 18 months
Reporting Status: Not Posted

8. Secondary Outcome: Cost Analysis (Self-reported)
Description: EuroQol five-dimensional (EQ-5D)
Time Frame: Baseline, 6 months, 13 months, and 18 months
Reporting Status: Not Posted

9. Secondary Outcome: Diabetes Emotional Distress (Self-reported)
Description: Problem Areas in Diabetes (PAID)
Time Frame: Baseline, 6 months, 13 months, and 18 months
Reporting Status: Not Posted

10. Secondary Outcome: Household Chaos (Self-reported)
Description: Confusion, Hubbub, and Order Scale (CHAOS)
Time Frame: Baseline, 6 months, 13 months, and 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Arm/Group | Standard Educational Care Control | The 3Ms Intervention + Standard Educational Care
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 29/74 | 24/75
Other Adverse Events (participants affected / at risk) | 29/74 | 21/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Educational Care Control (N=74) | The 3Ms Intervention + Standard Educational Care (N=75)
Diabetic ketoacidosis (Endocrine disorders) | 14 (22) | 11 (17)
New Non-diabetes-Related Health Problem (Surgical and medical procedures) | 2 (2) | 3 (4)
Blood glucose less than 50 mg/dL (Endocrine disorders) | 12 (16) | 10 (10)
Worsening Diabetes-Related Health Problem (Endocrine disorders) | 10 (14) | 6 (6)
New Psychiatric Problem (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Educational Care Control (N=74) | The 3Ms Intervention + Standard Educational Care (N=75)
Domestic violence (Social circumstances) | 1 (1) | 0 (0)
New Diabetes-Related Health Problem (Endocrine disorders) | 9 (9) | 5 (5)
New Non-diabetes-Related Health Problem (Surgical and medical procedures) | 16 (21) | 8 (12)
Problem with Parent-Child Relations (Social circumstances) | 1 (1) | 3 (3)
Psychiatric Problem (Psychiatric disorders) | 4 (4) | 4 (4)
School Related Problem (Social circumstances) | 4 (4) | 1 (1)
Worsening Diabetes-Related Health Problem (Endocrine disorders) | 7 (7) | 6 (7)
New Family Problem (Social circumstances) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03168867/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT03168867/ICF_001.pdf